CLINICAL TRIAL: NCT06304558
Title: "Effectiveness of Non-invasive Neuromodulation Treatment (NESA) for Improving Sexual Satisfaction in Healthy Subjects.
Brief Title: "Effectiveness of Non-invasive Neuromodulation Treatment for Improving Sexual Satisfaction in Healthy Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Vanesa Abuín, Associated Professor, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CI 240228, 2024-480
Record Dates: First submitted 2024-02-19; First posted 2024-03-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Sexual Satisfaction
MeSH Terms: conditions — Orgasm

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The Placebo group will mimic the Intervention group, but the device will not be connected. With this non-invasive neuromodulation, patiens do not experiment any sensation when the device is connected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): T The total number of sessions to be conducted for each patient will be 10 sessions, spread over 5 weeks, which means a frequency of twice a week.
  Each NESA microcurrent session will last 60 minutes. A maximum time of 15 minutes will be allowed for connecting the patient at the beginning and for removing the device at the end.
  During the 10 sessions of the treatment, the programming will evolve to optimize the response.
  The directing electrode will be located throughout the treatment between the spinous processes of C6 and C7 to act generally on the individual, and in later sessions, the electrode will be placed in the abdominal area to cover the hypogastric plexus and at S2-S3 to influence the sacral plexus.
  The intensity will be set to Low (3 volts) in all sessions, following the Arndt-Schulz law. The other device parameters range between 100-900 microamperes and between 1.14 and 14.29 hertz, and are preset by each program
  Interventions: Device: Non-Invasive Neuromodulation (NESA)
- Placebo (Placebo Comparator): Non-active Non-invasive Neuromodulation (NESA)
  Interventions: Device: Non-Invasive Neuromodulation (NESA)

INTERVENTIONS:
Device: Non-Invasive Neuromodulation (NESA) — Considering the objectives set: In the first phase, the directing electrode will be located at C6-C7 to generate a systemic and general effect on the organism, with program 1, program 2, program 7, and program 8. In the second phase, the directing electrode will be placed at the abdominal level in the area of the mesenteric plexus to influence the sympathetic innervation of the viscera. In the third phase, the directing electrode is located at S2-S3 to concentrate the action of the therapy on the sacral parasympathetic plexus,. In this way, both the sympathetic and parasympathetic innervation of the main sexual organs are covered through the sympathetic paravertebral ganglia and the sacral plexus.

SUMMARY:
The main objectives of the programming with the XSignal device will be to influence the sexual satisfaction of the participants.

As secondary objectives, the effectiveness of the XSignal device during a defined treatment period will be analyzed in terms of quality of life, pain, stress, anxiety, sexual function, sleep quality, cortisol, heart rate, blood pressure, respiratory rate, and body temperature of the same subjects, compared with a placebo group, observing the long-term influence of the results.

DETAILED DESCRIPTION:
Considering the objectives set: In the first phase, the directing electrode will be located at C6-C7 to generate a systemic and general effect on the organism, with program 1, program 2, program 7, and program 8. In the second phase, the directing electrode will be placed at the abdominal level in the area of the mesenteric plexus to influence the sympathetic innervation of the viscera. In the third phase, the directing electrode is located at S2-S3 to concentrate the action of the therapy on the sacral parasympathetic plexus,. In this way, both the sympathetic and parasympathetic innervation of the main sexual organs are covered through the sympathetic paravertebral ganglia and the sacral plexus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from 18 to 65 years
* Sexually active
* Signed consent form

Exclusion Criteria:

* Diagnosed diseases.
* Severe previous psychiatric conditions.
* Medical contraindications that prevent the use of non-invasive neuromodulation therapy.
* Having exercised in the hours prior to the NESA treatment.
* Having consumed coffee or tobacco in the hours prior to the treatment.
* Minors.
* Individuals who have previously received any type of neuromodulation treatment.
* Cancer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Sexual satisfaction | 10 minutes
  Questionnaire

SECONDARY OUTCOMES:
Stress levels | 10 minutes
  Questionnaire
Blood Pressure (Sistolic and diastolic) | 5 minutes
  Sfignomanometer
Heartbeats per minute | 5 minutes
  We Cardio http://en.wecardio.com/3_1ourmachinepage.html
Sleep Quality | 10 minutes
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrod, Villaviciosa de Odón, Spain

IPD SHARING:
Plan to Share IPD: No